CLINICAL TRIAL: NCT03136146
Title: Lead-In and Phase II Study of Clofarabine, Etoposide, Cyclophosphamide [CEC], Liposomal Vincristine (VCR), Dexamethasone and Bortezomib in Relapsed/Refractory Acute Lymphoblastic Leukemia (ALL) and Lymphoblastic Lymphoma (LL)
Brief Title: Combination Chemotherapy in Treating Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia, Lymphoblastic Lymphoma, Burkitt Lymphoma/Leukemia, or Double-Hit Lymphoma/Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0211; NCI-2018-01198 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0211 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Acute Lymphoblastic Leukemia; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Burkitt Leukemia; Recurrent Burkitt Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Refractory Acute Lymphoblastic Leukemia; Refractory Burkitt Leukemia; Refractory Burkitt Lymphoma; Refractory High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Refractory Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Bortezomib; Clofarabine; Cyclophosphamide; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Etoposide; ofatumumab; pegfilgrastim; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): See detailed description
  Interventions: Drug: Bortezomib; Drug: Clofarabine; Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Etoposide; Biological: Ofatumumab; Biological: Pegfilgrastim; Biological: Rituximab; Drug: Vincristine Sulfate Liposome

INTERVENTIONS:
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Clofarabine — Given IV
  Other Names: Clofarex; Clolar
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Biological: Ofatumumab — Given IV
  Other Names: Arzerra; GSK1841157; HuMax-CD20; HuMax-CD20, 2F2; Kesimpta
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; filgrastim-SD/01; Fulphila; HSP-130; Jinyouli; Neulasta; Neulastim; Nyvepria; PEG-filgrastim; Pegcyte; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Nyvepria; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim Biosimilar Udenyca; Pegfilgrastim Biosimilar Ziextenzo; pegfilgrastim-apgf; pegfilgrastim-bmez; pegfilgrastim-cbqv; Pegfilgrastim-jmdb; SD-01; SD-01 sustained duration G-CSF; Udenyca; Ziextenzo
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima
Drug: Vincristine Sulfate Liposome — Given IV
  Other Names: Marqibo

SUMMARY:
This phase II trial studies the side effects and how well combination chemotherapy works in treating patients with acute lymphoblastic leukemia, lymphoblastic lymphoma, Burkitt lymphoma/leukemia, or double-hit lymphoma/leukemia that has come back or does not respond to treatment. Drugs used in chemotherapy, such as clofarabine, etoposide, cyclophosphamide, vincristine sulfate liposome, dexamethasone and bortezomib, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To collect the safety/toxicity information and assess the initial efficacy information (objective overall response rate: complete response [CR]+ CR with incomplete platelet recovery [CRp]/CR with incomplete bone marrow recovery [CRi]) after treatment with clofarabine, etoposide, cyclophosphamide (CEC), vincristine sulfate liposome (liposomal vincristine) (VCR), dexamethasone and bortezomib in relapsed/refractory acute lymphoblastic leukemia (ALL) or lymphoblastic lymphoma (LL) including relapsed/refractory Philadelphia (Ph) positive B-ALL/LL or Burkitt's leukemia/lymphoma or double-hit leukemia/lymphoma.

SECONDARY OBJECTIVE:

I. To determine the CR duration, event free survival (EFS), and overall survival (OS) after treatment with CEC, liposomal VCR, dexamethasone and bortezomib in relapsed/refractory ALL or LL including relapsed/refractory Ph positive B-ALL/LL or Burkitt's leukemia/lymphoma or double-hit leukemia/lymphoma.

OUTLINE:

INDUCTION: Patients receive clofarabine intravenously (IV) over 1-2 hours on days 1-5, etoposide IV over 2 hours on days 1-5, cyclophosphamide IV over 1 hour on days 1-5, vincristine sulfate liposome IV over 1 hour on days 2 and 11, dexamethasone orally (PO) daily or IV over 15 minutes on days 1-5, bortezomib subcutaneously (SC) on days 1, 4, 8 and 11, ofatumumab or rituximab IV over 4-24 hours on days 2 and 11, and pegfilgrastim SC on day 6 in the absence of disease progression or unacceptable toxicity. Patients may receive 1 additional course of induction therapy depending on the disease response.

CONSOLIDATION THERAPY: Patients receive clofarabine IV over 1-2 hours on days 1-4, etoposide IV over 2 hours on days 1-4, cyclophosphamide IV over 1 hour on days 1-4, vincristine sulfate liposome IV over 1 hour on days 2 and 11, dexamethasone PO or IV over 15 minutes on days 1-5, bortezomib SC on days 1, 4, 8 and 11, pegfilgrastim SC on day 6. Treatment repeats every 28 days for up to 5 courses in the absence of disease progression or unacceptable toxicity. Patients may receive ofatumumab or rituximab IV over 4-24 hours on days 2 and 11 for 4 courses.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/refractory acute lymphoblastic leukemia (ALL) or lymphoblastic lymphoma (LL):

  * Relapsed and/or refractory Philadelphia negative acute lymphoblastic leukemia or lymphoblastic lymphoma (LL) (Lead-in and Phase II)
  * Relapsed and/or refractory Philadelphia positive acute lymphoblastic leukemia, Burkitt leukemia/lymphoma or "double-hit" leukemia/lymphoma (phase II only)
* At least 21 days elapsed from prior systemic chemotherapy (at least 14 days elapsed from prior systemic chemotherapy in the setting of rapidly progressive disease without significant residual extramedullary toxicity). Hydroxyurea and dexamethasone permitted up to approximately 24 hours prior to the start of therapy. Interruption of tyrosine kinase inhibitor (TKI) not required in Ph positive ALL subset
* Age older than 15 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 3 (There may be certain patients with performance status [PS] 3 in the context of rapidly proliferative/refractory ALL who would benefit from this regimen. We don't want to exclude such patients who may derive benefit from this salvage regimen)
* Serum bilirubin =< 1.5 mg/dL
* Serum glutamate pyruvate transaminase (SGPT) =< 3 x upper limit normal (ULN), with exception for Gilbert's syndrome
* Estimated creatinine clearance or GFR (glomerular filtration rate) >= 50 mL/min
* Signed informed consent

Exclusion Criteria:

* Active >= grade 3 peripheral neuropathy
* Active hepatic graft-versus-host disease
* Known positivity for hepatitis B or C
* Pregnancy
* Breast feeding

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-08-09 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 8 years
  The severity of the toxicities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events.
Overall response rate (ORR) (Phase II) | Up to 8 years
  Will be estimated along with the exact 95% confidence interval.

SECONDARY OUTCOMES:
Overall survival | From initiation of treatment, assessed up to 8 years
  Will be estimated using the method of Kaplan and Meier. The log-rank tests will be used to compare the time-to-event outcomes among subgroups of patients.
Event free survival | From the treatment start, assessed up to 8 years
  Will be estimated using the method of Kaplan and Meier. The log-rank tests will be used to compare the time-to-event outcomes among subgroups of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Maro Ohanian, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org